CLINICAL TRIAL: NCT06158906
Title: Validity of Web-Based OSDI-6 Questionnaire in a Chinese Adult Population
Status: Completed | Type: Observational
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: OSDI6
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-11

CONDITIONS: Dry Eye
Keywords: qestionnaire
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Dry eye patients were recruited to fill in the questionnaire

SUMMARY:
This study aimed to evaluate the validity of the Chinese translation version of OSDI-6 (C-OSDI-6) in a theoretical set-up of two questionnaire groups for dry eye

DETAILED DESCRIPTION:
Screening for dry eye symptoms and quantifying dry eye symptoms aids in assessment, diagnosis, and treatment. Patient-reported outcome (PRO) instruments such as the Ocular Surface Disease Index (OSDI-12) are utilized for assessing patients' subjective experiences and functional abilities. The OSDI-12 comprises of 12-item and is often used in conjunction with other tests in clinical settings to assess individuals with DE. Created in 1997, the original OSDI consisted of 12 items and was designed to evaluate subjective dry eye symptoms and the consequences of DED on vision-related activities of daily life over the preceding week. The 12 items are grouped into three subscales: ocular symptoms (three items), vision-related functions (six items), and environmental triggers (three items). While the original version of the OSDI-12 questionnaire was created in English and was later translated and validated into other languages, it should be used carefully since the cutoff values vary among various languages (27.2 points for the Chinese version and 36.3 points for the Japanese version) . Recent research using Rasch analysis found that separating answer items into four categories by merging "half of the time" and "most of the time" might lead to higher thresholds and better intervals in each category. The OSDI-12 total score is calculated using the formula: [(sum of scores for all questions answered) × 100]/ [(total number of questions answered) × 4]. Ocular Surface Disease Index-6 (OSDI-6) is a derivative and shortened version of the original OSDI-12 and can potentially improve efficiency in a busy clinical setting.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed dry eye
* Able and willing to comply with the schedule
* Able to read and understand the C-OSDI-12 questionnaire independently

Exclusion Criteria:

* The researchers judged to be not suitable

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed with dry eye
Sampling Method: Probability Sample
Enrollment: 270 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-02-17 (Actual); Study Completion 2024-02-17 (Actual)

PRIMARY OUTCOMES:
OSDI12 | Baseline
  The patient will answer each question on a scale ranging from 0 to 4, with 0 indicating 'none of the time' and 4 indicating 'all of the time'. If a certain question is deemed irrelevant, it will be marked as 'not applicable (N/A)' and excluded from the analysis. The OSDI total score is calculated according to the following formula. The scale ranges from 0 to 100, with higher scores representing more severe cases of dry eye syndrome

CONTACTS AND LOCATIONS:
Locations (1):
- He Eye Hospital, Shenyang, None Selected, China

REFERENCES:
- [Background] Jones L, Downie LE, Korb D, Benitez-Del-Castillo JM, Dana R, Deng SX, Dong PN, Geerling G, Hida RY, Liu Y, Seo KY, Tauber J, Wakamatsu TH, Xu J, Wolffsohn JS, Craig JP. TFOS DEWS II Management and Therapy Report. Ocul Surf. 2017 Jul;15(3):575-628. doi: 10.1016/j.jtos.2017.05.006. Epub 2017 Jul 20. PMID 28736343
- [Background] Craig JP, Nichols KK, Akpek EK, Caffery B, Dua HS, Joo CK, Liu Z, Nelson JD, Nichols JJ, Tsubota K, Stapleton F. TFOS DEWS II Definition and Classification Report. Ocul Surf. 2017 Jul;15(3):276-283. doi: 10.1016/j.jtos.2017.05.008. Epub 2017 Jul 20. PMID 28736335
- [Background] Schiffman RM, Christianson MD, Jacobsen G, Hirsch JD, Reis BL. Reliability and validity of the Ocular Surface Disease Index. Arch Ophthalmol. 2000 May;118(5):615-21. doi: 10.1001/archopht.118.5.615. PMID 10815152
- [Background] Nichols KK, Mitchell GL, Zadnik K. Performance and repeatability of the NEI-VFQ-25 in patients with dry eye. Cornea. 2002 Aug;21(6):578-83. doi: 10.1097/00003226-200208000-00009. PMID 12131034
- [Background] Lu F, Tao A, Hu Y, Tao W, Lu P. Evaluation of Reliability and Validity of Three Common Dry Eye Questionnaires in Chinese. J Ophthalmol. 2018 Aug 27;2018:2401213. doi: 10.1155/2018/2401213. eCollection 2018. PMID 30225139
- [Background] Midorikawa-Inomata A, Inomata T, Nojiri S, Nakamura M, Iwagami M, Fujimoto K, Okumura Y, Iwata N, Eguchi A, Hasegawa H, Kinouchi H, Murakami A, Kobayashi H. Reliability and validity of the Japanese version of the Ocular Surface Disease Index for dry eye disease. BMJ Open. 2019 Nov 25;9(11):e033940. doi: 10.1136/bmjopen-2019-033940. PMID 31772113